CLINICAL TRIAL: NCT05361304
Title: Clinical Evaluation of Senofilcon A Contact Lenses Using a Novel Manufacturing Technology
Brief Title: Clinical Evaluation of Senofilcon A Contact Lenses Using a Novel Manufacturing Technology to Evaluate Overall Visual Acuity.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR-6474
Record Dates: First submitted 2022-04-29; First posted 2022-05-04 (Actual); Results first posted 2023-07-13 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-06

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- TEST Lens (Experimental): Eligible subjects who are habitual soft contact lens wearers will be randomized into the TEST Lens for the duration of the study.
  Interventions: Device: senofilcon A contact lenses made with a novel manufacturing technology
- CONTROL Lens (Experimental): Eligible subjects who are habitual soft contact lens wearers will be randomized into the CONTROL Lens for the duration of the study.
  Interventions: Device: senofilcon A contact lenses made with the current manufacturing technology

INTERVENTIONS:
Device: senofilcon A contact lenses made with a novel manufacturing technology — TEST Lens
  Arms: TEST Lens
Device: senofilcon A contact lenses made with the current manufacturing technology — CONTROL Lens
  Arms: CONTROL Lens

SUMMARY:
This study is a feasibility, multi-site, randomized, double-masked, 2-arm parallel group design, 2-week dispensing study with weekly visits to evaluate visual acuity.

ELIGIBILITY:
Inclusion Criteria:

Potential subjects must satisfy all of the following criteria to be enrolled in the study:

1. Read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
3. Be between 18 and 39 (inclusive) years of age at the time of screening.
4. By self-report, habitually wear spherical soft silicone hydrogel contact lenses in both eyes in a daily reusable or daily disposable wear modality (i.e. not extended wear modality). Habitual wear is defined as a minimum of 6 hours of wear per day, for a minimum of 5 days per week during the past 30 days.
5. Possess a wearable pair of spectacles that provide correction for distance vision.
6. The spherical equivalent of the subject's vertex-corrected distance refraction must be between -1.00 and -6.00 DS (inclusive) in each eye.
7. The magnitude of the cylindrical component of the subject's vertex-corrected distance refraction must be between 0.00 and 1.00 DC (inclusive) in each eye.
8. The best corrected, monocular, distance visual acuity must be 20/25 or better in each eye.

Exclusion Criteria:

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

1. Be currently pregnant or lactating.
2. Be currently using any ocular medications or have any ocular infection of any type.
3. By self-report, have any ocular or systemic disease, allergies, infection, or use of medication that the investigator believes might contraindicate or interfere with contact lens wear, or otherwise compromise study endpoints, including infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive disease (e.g., Human Immunodeficiency Virus [HIV]), autoimmune disease (e.g. rheumatoid arthritis, Sjögren's syndrome), or history of serious mental illness or seizures. See section 9.1 for additional details regarding excluded systemic medications.
4. Be currently wearing monovision or multifocal contact lenses.
5. Be currently wearing lenses in an extended wear modality.
6. Have participated in a contact lens or lens care product clinical trial within 7 days prior to study enrollment.
7. Be an employee (e.g., Investigator, Coordinator, Technician) or immediate family member of an employee (including partner, child, parent, grandparent, grandchild or sibling of the employee or their spouse) of the clinical site.
8. Have clinically significant (grade 3 or higher on the FDA grading scale) slit lamp findings (e.g., corneal edema, neovascularization or staining, tarsal abnormalities or bulbar injection) or other corneal or ocular disease or abnormalities that the investigator believes will contraindicate contact lens wear or may otherwise compromise study endpoints (including entropion, ectropion, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, moderate or above corneal distortion, herpetic keratitis). (Specify method of determination if needed).
9. Have fluctuations in vision due to clinically significant dry eye or other ocular conditions.
10. Have had or have planned (within the study period) any ocular or intraocular surgery (e.g., radial keratotomy, PRK, LASIK, iridotomy, retinal laser photocoagulation, etc.).

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 123 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2022-07-05 (Actual); Study Completion 2022-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care, Inc. Clinical Trial, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (6):
- United States (6):
  - VRC, Jacksonville, Florida
  - Flora Chen Poveda OD, PA - Orange Park, Orange Park, Florida
  - Tallahassee Eye Center, Tallahassee, Florida
  - Sacco Eye Group, Vestal, New York
  - William J. Bogus, O.D., Salt Lake City, Utah
  - Botetourt Eyecare, LLC, Salem, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 123 subjects were enrolled in this study. Of those enrolled, all 123 subjects were dispensed at least one study lens. Of those dispensed, 118 subjects completed the study while 5 subjects were discontinued.
Groups:
- Senofilcon A Contact Lenses Made With the Current Manufacturing Technology: Subjects that wore the Senofilcon A contact lenses made with the current manufacturing technology lens during the study.
- Senofilcon A Contact Lenses Made With a Novel Manufacturing Technology: Subjects that wore the Senofilcon A contact lenses made with a novel manufacturing technology lens during the study.
Period: Overall Study
Arm/Group | Senofilcon A Contact Lenses Made With the Current Manufacturing Technology | Senofilcon A Contact Lenses Made With a Novel Manufacturing Technology
Started | 62 | 61
Completed | 59 | 59
Not Completed | 3 | 2
Not completed — Senofilcon A contact lenses made with a novel manufacturing technology Article Not Available. | 1 | 0
Not completed — COVID-19 Related | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: All subjects dispensed a study lens
Groups:
- Total: Total of all reporting groups
Arm/Group | Senofilcon A Contact Lenses Made With the Current Manufacturing Technology | Senofilcon A Contact Lenses Made With a Novel Manufacturing Technology | Total
Number analyzed (Participants) | 62 | 61 | 123
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.1 (5) | 30.7 (5.85) | 30.4 (5.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 42 | 90
  Male | 14 | 19 | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 2 | 4
  Black or African American | 8 | 6 | 14
  White | 52 | 52 | 104
  Multiple | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States: participants | 62 | 61 | 123

OUTCOME MEASURES:

1. Primary Outcome: Monocular logMAR Visual Acuity
Description: Monocular visual acuity was measured on a logMAR (Logarithm of Minimal Angle of Resolution) scale under high luminance low contrast (HLLC), and low luminance high contrast (LLHC) at distance (4 meters) using an ETDRS (Early Treatment Diabetic Retinopathy Study) charts. Letter-by-letter results calculated the visual performance score for each chart read. LogMAR scores closer to zero, or below zero, indicate a better visual acuity. A logMAR visual performance score of 0.0 is equivalent to Snellen visual acuity of 20/20.
Time Frame: 2-Week Follow-up
Population: All subjects who successfully completed all study visits without a major protocol deviation at 2-Week Follow-up evaluation.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Senofilcon A Contact Lenses Made With the Current Manufacturing Technology | Senofilcon A Contact Lenses Made With a Novel Manufacturing Technology
Number analyzed (Participants) | 59 | 59
Number analyzed (eyes) | 118 | 118
logMAR
  High Luminance Low Contrast | 0.051 (0.1082) | 0.032 (0.0947)
  Low Luminance High Contrast | 0.044 (0.1042) | 0.036 (0.0830)
Statistical Analysis 1: Comparison: Senofilcon A Contact Lenses Made With the Current Manufacturing Technology vs Senofilcon A Contact Lenses Made With a Novel Manufacturing Technology; It was calculated using a 2 independent sample means t-test with a 2-sided type I error rate of 5% with at least 80% statistical power, that 100 subjects were required to test for non-inferiority of the Senofilcon A contact lenses made with a novel manufacturing technology compared to the Senofilcon A contact lenses made with the current manufacturing technology for distance (4m) under HLLC; Test type: Non-Inferiority; Linear Mixed Model; Kenward and Roger method was used for denominator degrees of freedom; Least square Mean (LSM) Difference = -0.020, 95% CI 2-sided [-0.040 to 0.000], Standard Error of Mean 0.012 — LSM difference was calculated as Senofilcon A contact lenses made with a novel manufacturing technology minus Senofilcon A contact lenses made with the current manufacturing technology
Statistical Analysis 2: Comparison: Senofilcon A Contact Lenses Made With the Current Manufacturing Technology vs Senofilcon A Contact Lenses Made With a Novel Manufacturing Technology; It was calculated using a 2 independent sample means t-test with a 2-sided type I error rate of 5% with at least 80% statistical power, that 100 subjects were required to test for non-inferiority of the Senofilcon A contact lenses made with a novel manufacturing technology compared to the Senofilcon A contact lenses made with the current manufacturing technology for distance (4m) under LLHC; Test type: Non-Inferiority; Linear Mixed Model; Kenward and Roger method was used for denominator degrees of freedom; Least square Mean (LSM) Difference = -0.010, 95% CI 2-sided [-0.030 to 0.020], Standard Error of Mean 0.012 — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Average Daily Wearing Time
Description: Average daily wear time was assessed by calculating the number of hours between subjects reported time of insertion and time of removal of the study lenses, on an average day.
Time Frame: 2-Week Follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Senofilcon A Contact Lenses Made With a Novel Manufacturing Technology: Subjects randomized to receive the Senofilcon A contact lenses made with a novel manufacturing technology lens during the study
Arm/Group | Senofilcon A Contact Lenses Made With the Current Manufacturing Technology | Senofilcon A Contact Lenses Made With a Novel Manufacturing Technology
Number analyzed (Participants) | 59 | 59
hours | 14.2 (2.12) | 14.5 (1.97)
Statistical Analysis 1: Comparison: Senofilcon A Contact Lenses Made With the Current Manufacturing Technology vs Senofilcon A Contact Lenses Made With a Novel Manufacturing Technology; It was calculated using a 2 independent sample means t-test with a 2-sided type I error rate of 5% with at least 80% statistical power, that 100 subjects were required to test for non-inferiority of the Senofilcon A contact lenses made with a novel manufacturing technology compared to the Senofilcon A contact lenses made with the current manufacturing technology; Test type: Non-Inferiority; Linear Mixed Model; Kenward and Roger method was used for denominator degrees of freedom; Least square Mean (LSM) Difference = 0.270, 95% CI 2-sided [-0.460 to 1.010], Standard Error of Mean 0.370 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: CLUE Comfort Score
Description: Subjective vision was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120. The average CLUE comfort score for each lens type was reported.
Time Frame: 2-Week Follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Senofilcon A Contact Lenses Made With the Current Manufacturing Technology | Senofilcon A Contact Lenses Made With a Novel Manufacturing Technology
Number analyzed (Participants) | 59 | 59
Units on a scale | 71.53 (28.439) | 76.06 (21.838)
Statistical Analysis 1: Comparison: Senofilcon A Contact Lenses Made With the Current Manufacturing Technology vs Senofilcon A Contact Lenses Made With a Novel Manufacturing Technology; Test type: Non-Inferiority; Linear Mixed Model; Kenward and Roger method was used for denominator degrees of freedom; LSM Difference = 4.0, 95% CI 2-sided [-4.1 to 12.0], Standard Error of Mean 4.06 — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: CLUE Vision Score
Description: Subjective vision was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120. The average CLUE vision score for each lens type was reported.
Time Frame: 2-Week Follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Senofilcon A Contact Lenses Made With the Current Manufacturing Technology: Subjects randomized to receive the Senofilcon A contact lenses made with the current manufacturing technology lens during the study
Arm/Group | Senofilcon A Contact Lenses Made With the Current Manufacturing Technology | Senofilcon A Contact Lenses Made With a Novel Manufacturing Technology
Number analyzed (Participants) | 59 | 59
Units on a scale | 73.28 (24.077) | 74.26 (20.615)
Statistical Analysis 1: Comparison: Senofilcon A Contact Lenses Made With the Current Manufacturing Technology vs Senofilcon A Contact Lenses Made With a Novel Manufacturing Technology; Test type: Non-Inferiority — Non-inferiority was declared if the lower bound of the confidence interval of the mean difference between Senofilcon A contact lenses made with a novel manufacturing technology and Senofilcon A contact lenses made with the current manufacturing technology is greater than -5; Linear Mixed Model; Kenward and Roger method was used for denominator degrees of freedom; LSM Differences = -0.3, 95% CI 2-sided [-7.1 to 6.5], Standard Error of Mean 3.44 — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study; The study duration for each subject was approximately 2 weeks.
Description: All subjects dispensed a study lens.
Arm/Group | Senofilcon A Contact Lenses Made With the Current Manufacturing Technology | Senofilcon A Contact Lenses Made With a Novel Manufacturing Technology
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/61
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/61
Other Adverse Events (participants affected / at risk) | 0/62 | 0/61

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-19): https://cdn.clinicaltrials.gov/large-docs/04/NCT05361304/Prot_SAP_000.pdf